CLINICAL TRIAL: NCT03707548
Title: A Clinical Trial of Group-based Body Psychotherapy (BPT) to Improve Bodily Disturbances in Post-treatment Cancer Patients in Combination With Randomized Controlled Smartphone-triggered Bodily Interventions
Brief Title: BPT to Improve Bodily Disturbances in Post-treatment Cancer Patients
Acronym: KPTK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-01115; me17Schaefert2
Record Dates: First submitted 2018-09-26; First posted 2018-10-16 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Cancer Patients
Keywords: body psychotherapy; smartphone-triggered interventions; psychosocial impairments related to cancer; cancer-related disturbances in bodily wellbeing; Body Image Scale; group psychotherapy; bodily disturbances in post-treatment cancer patients

STUDY DESIGN:
Intervention Model Description: Study design: The project follows the outline of a non-randomized evaluation of a weekly group BPT using a waiting-period comparator, with a nested randomized controlled trial (RCT) to evaluate the short-term efficacy of smartphone-triggered bodily interventions.
  Measurement points:
  * Patients will be surveyed at three points in time (initial consultation, pre- and post-intervention) to explore the effects of BPT on bodily disturbances and body image in post-treatment cancer patients.
  * During the BPT Intervention group cohesion and bodily well-being will be assessed weekly.
  * The smartphone-triggered bodily and control interventions will be provided over a period of 5 consecutive weeks on 6 days per week and will be assessed pre- and post intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group BPT (Experimental): Six group BPT sessions (using a waiting-period comparator and pre-/post design)
  A nested randomized controlled trial (RCT) is included to evaluate the short-term efficacy of smartphone-triggered bodily interventions compared with the smartphone triggered control intervention of audio-typed fairy tales.
  Interventions: Behavioral: BPT; Behavioral: Smartphone-triggered bodily interventions; Behavioral: Smartphone triggered control intervention

INTERVENTIONS:
Behavioral: BPT — BPT will consist of 6 weekly group sessions, based on a scientific approach, integrating body-oriented techniques to improve patients' awareness, perception, acceptance, and expression regarding their body.
Behavioral: Smartphone-triggered bodily interventions — Smartphone-triggered bodily interventions will consist of brief BPT exercises insuring the transfer from the group BPT sessions into patients' daily lives. Smartphone bodily interventions will be triggered by short audio-clips.
Behavioral: Smartphone triggered control intervention — The smartphone triggered control intervention will be selected fairy tales presented by audio-clips.

SUMMARY:
With this project investigators focus on the evaluation whether bodily disturbances in post-treatment cancer patients can be influenced positively by group BPT and if intermittent smartphone-triggered bodily interventions are effective.

DETAILED DESCRIPTION:
Background: Disturbances in bodily wellbeing represent one key aspect of psychosocial impairments related to cancer. Therefore, interventions to improve bodily wellbeing in post-treatment cancer patients are important.

Objectives: This project aims at two goals:

1. Investigators want to evaluate whether bodily disturbances in post-treatment cancer patients can be influenced positively by group BPT (Non-randomized evaluation of a weekly group BPT using a waiting-period comparator).
2. In addition the efficacy of intermittent smartphone-triggered bodily interventions is assessed with a nested RCT to evaluate short-term efficacy of smartphone-triggered bodily interventions.

Study design: The project follows the outline of a non-randomized evaluation of a weekly group BPT using a waiting-period comparator, with a nested randomized controlled trial (RCT) to evaluate the short-term efficacy of smartphone-triggered bodily interventions.

Study flow:

* Participants will first undergo a waiting period (duration at least 6 weeks) followed by the group BPT (6 weekly sessions, 90 minutes each).
* During the group BPT, either a smartphone-triggered bodily intervention or a smartphone-triggered control intervention will be provided at random (randomization on a daily basis) over a period of 5 consecutive weeks on 6 days per week. This will result in 15 smartphone-triggered bodily interventions and 15 smartphone-triggered control interventions, which each patient will undergo.

Measurement points: Patients will be surveyed at three points in time (initial consultation, pre- and post-intervention). Standardized questionnaires will be used to measure patients' body disturbances, body image, body mindfulness, physical complaints, quality of life, vitality, mental health, anxiety and depression and to explore the effects of BPT on bodily disturbances and body image in post-treatment cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Having received curatively intended treatment for any malignant neoplasm; primary treatment (surgery, radiotherapy, chemotherapy) being completed >/= 3 months ago before study inclusion. Any other ongoing anti-tumor therapy is allowed (e.g., hormonal therapy, adjuvant immunotherapy)
* existing bodily disturbances
* No sign of progress or recurrence of malignancy at study inclusion according to treating physician
* Score of 0 or 1 according to the Eastern Cooperative Oncology Group (ECOG) Performance Score
* Having an anticipated life expectancy of >/= 12 months, according to treating physician
* age 18 years or older
* Capacity to participate in group BPT sessions in Basel or Winterthur, 3 study assessments, and the smartphone-triggered interventions
* Ability to provide informed consent

Exclusion Criteria:

* Suffering from a severe current mental disorder
* Risk of current suicidality, as indicated by a suicide item score >/= 2 in the BDI-II (Beck Depression Inventory), as this group BPT intervention is not appropriate to support suicidal patients in acute crises
* Participation in any other clinical trial with a psychosocial intervention
* Receiving any other current psychotherapeutic treatment with the exception of already established therapies
* Inability to understand and speak German

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
Changes in bodily disturbances assessed by questionnaires | Questionnaire at baseline and 6 weeks after baseline (=after the waiting period;pre-therapy) and 14 weeks after baseline (=post-therapy)
  self-perception of change in appearance and displeasure with change or perceived change in appearance; assessed via Body Image Scale (BIS). BIS total score is calculated by adding the score obtained on each item, yielding a possible range from 0-30. Higher scores indicate a higher degree of body image dissatisfaction.

SECONDARY OUTCOMES:
Changes in bodily wellbeing | applied twice on each training day of the smartphone-triggered interventions: first directly preceding, second directly following the smartphone-triggered interventions
  bodily wellbeing is assessed by Multidimensional Mood Questionnaire (MDMQ). 3 scales are calculated: "good-bad", and "awake-tired", "calm-nervous". Scores are calculated by adding the score obtained on each item, yielding a possible range from 4-20 in each scale. Higher values represent a better outcome.
Changes in mood | applied twice on each training day of the smartphone-triggered interventions: first directly preceding, second directly following the smartphone-triggered interventions
  mood is assessed by Multidimensional Mood Questionnaire (MDMQ). 3 scales are calculated: "good-bad", and "awake-tired", "calm-nervous". Scores are calculated by adding the score obtained on each item, yielding a possible range from 4-20 in each scale. Higher values represent a better outcome.
Changes in body mindfulness | Questionnaire at baseline and 6 weeks after baseline (=after the waiting period;pre-therapy) and 14 weeks after baseline (=post-therapy)
  assessed by Body Mindfulness Questionnaire (BMQ). 2 scales are calculated: "Experiencing Body Awareness", and "Appreciating Body Awareness". Scores are calculated by adding the score obtained on each item, yielding a possible range from 7-42 in each scale. Higher values represent a better outcome.
Changes in somatic symptoms | Questionnaire at baseline and 6 weeks after baseline (=after the waiting period;pre-therapy) and 14 weeks after baseline (=post-therapy)
  somatic symptoms are assessed by the EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 items). All scales and single-item measures range in scores from 0 to 100. A high score represents a high level of symptomatology. The following somatic symptom scales are calculated: fatigue, nausea and vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhoea. The principle for scoring these scales is the same in all cases: 1.The average of the items that contribute to the scale is estimated; this is the raw score. 2. A linear transformation is used to standardise the raw score, so that scores range from 0 to 100.
Changes in somatic symptom disorder-B criteria | Questionnaire at baseline and 6 weeks after baseline (=after the waiting period;pre-therapy) and 14 weeks after baseline (=post-therapy)
  somatic symptom disorder-B criteria are assessed by Somatic Symptom Disorder-B Criteria Scale (SSD-12). 1 total score and 3 subscores are calculated: "cognitive aspects", "affective aspects", and "behavioral aspects". Scores are calculated by adding the score obtained on each item. Range for subscales: 0-16; range for total score: 0-48; higher scores are representing greater severity.
Changes in distress | Questionnaire at baseline and 6 weeks after baseline (=after the waiting period;pre-therapy) and 14 weeks after baseline (=post-therapy)
  distress is assessed by National Comprehensive Cancer Network Distress Thermometer (DT). A visual analogue scale ranging from 0=no distress to 10=extreme distress.
Changes in anxiety | Questionnaire at baseline and 6 weeks after baseline (=after the waiting period;pre-therapy) and 14 weeks after baseline (=post-therapy)
  anxiety is assessed by the anxiety subscale of the Hospital Anxiety and Depression Scale (HADS-A). The anxiety-score is calculated by adding the score obtained on each item, range 0-21, with higher scores representing greater severity.
Changes in depression | Questionnaire at baseline and 6 weeks after baseline (=after the waiting period;pre-therapy) and 14 weeks after baseline (=post-therapy)
  Depression is assessed by the depression subscale of the Hospital Anxiety and Depression Scale (HADS-D). The depression-score is calculated by adding the score obtained on each item, range 0-21, with higher scores representing greater severity.
Changes in vitality | Questionnaire at baseline and 6 weeks after baseline (=after the waiting period;pre-therapy) and 14 weeks after baseline (=post-therapy)
  vitality is assessed by the 36-Item Short Form Health Survey (SF-36) - scale vitality. Items in the scale are averaged together to create the vitality score. Range from 0 to 100, a higher score defining a more favorable health state.
Changes in mental health | Questionnaire at baseline and 6 weeks after baseline (=after the waiting period;pre-therapy) and 14 weeks after baseline (=post-therapy)
  mental health is assessed by the 36-Item Short Form Health Survey (SF-36) - scale mental health. Items in the scale are averaged together to create the mental health score. Range from 0 to 100, a higher score defining a more favorable health state.
Changes in quality of life | Questionnaire at baseline and 6 weeks after baseline (=after the waiting period;pre-therapy) and 14 weeks after baseline (=post-therapy)
  quality of life is assessed by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 items (EORTC QLQ-C30). The following scales are computed: global health status/quality of life, physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning. All scales range in scores from 0 to 100. A high score for a functional scale represents a high level of functioning, a high score for the global health status represents a high quality of life. The principle for scoring these scales is the same in all cases: 1.The average of the items that contribute to the scale is estimated; this is the raw score. 2. A linear transformation is used to standardise the raw score, so that scores range from 0 to 100.
Changes in suicidal tendency | Questionnaire at baseline and 6 weeks after baseline (=after the waiting period;pre-therapy) and 14 weeks after baseline (=post-therapy)
  suicidal tendency is assessed by the Beck Depression Inventory (BDI-II), Item I: Suicidal tendency. Range from 0 to 3, a higher value representing a higher suicidal tendency.

OTHER OUTCOMES:
Changes in bodily disturbances assessed by semistructured interview | qualitative assessment at baseline and 14 weeks after baseline (=post-therapy)
  self-perception of change in appearance and displeasure with change or perceived change in appearance; assessed via semistructured interview
Change in group cohesion | assessed 7, 8, 9, 10, 11 and 12 weeks after baseline directly after each group session
  Group cohesion is assessed by the Group Climate Questionnaire - Short Form (GCQ-S). The questionnaire consists of a total score and 3 subscales (all ranges from 0 to 6): Scale 1: Engaged: This describes the positive working group atmosphere. Scale 2: Conflict: This reflects anger and tension in the group. Scale 3: Avoiding: This describes behaviors indicating avoidance of personal responsibility of group work by the members. Higher values represent a higher degree in engagement, conflict, or avoiding. Scales scores are determined by calculating the mean of the relevant items.

CONTACTS AND LOCATIONS:
Overall Officials: Rainer M Schaefert, Prof. Dr. MD, Study Chair — Department of Psychosomatics/ Division of Medicine; Astrid Grossert, MSc, Principal Investigator — Department of Psychosomatics/ Division of Medicine
Locations (2):
- Switzerland (2):
  - Department of Psychosomatics/ Division of Medicine; University Hospital of Basel, Basel
  - Department of Oncology and Hematology; Kantonsspital Winterthur, Winterthur

REFERENCES:
- [Background] Grossert A, Meinlschmidt G, Schaefert R. A case series report of cancer patients undergoing group body psychotherapy. F1000Res. 2017 Sep 5;6:1646. doi: 10.12688/f1000research.12262.2. eCollection 2017. PMID 29067164
- [Derived] Meinlschmidt G, Grossert A, Meffert C, Roemmel N, Hess V, Rochlitz C, Pless M, Hunziker S, Wossmer B, Geuter U, Schaefert R. Smartphone-Based Psychotherapeutic Interventions in Blended Care of Cancer Survivors: Nested Randomized Clinical Trial. JMIR Cancer. 2023 Aug 28;9:e38515. doi: 10.2196/38515. PMID 37639296
- [Derived] Grossert A, Meffert C, Hess V, Rochlitz C, Pless M, Hunziker S, Wossmer B, Geuter U, Meinlschmidt G, Schaefert R. Group-based body psychotherapy improves appreciation of body awareness in post-treatment cancer patients: A non-randomized clinical trial. Front Psychol. 2023 Apr 6;14:956493. doi: 10.3389/fpsyg.2023.956493. eCollection 2023. PMID 37089722
- [Derived] Grossert A, Meffert C, Hess V, Rochlitz C, Pless M, Hunziker S, Wossmer B, Geuter U, Meinlschmidt G, Schaefert R. A clinical trial of group-based body psychotherapy to improve bodily disturbances in post-treatment cancer patients in combination with randomized controlled smartphone-triggered bodily interventions (KPTK): study protocol. BMC Psychol. 2019 Dec 30;7(1):90. doi: 10.1186/s40359-019-0357-1. PMID 31888741